CLINICAL TRIAL: NCT00176176
Title: Change of EEG Activity and Cerebral Circulation During Induced Ventricular Fibrillation and Investigation of Cognitive Function Before and After Induced Ventricular Fibrillation in EP Study
Brief Title: Investigation of Cognitive Function Before and After Induced Ventricular Fibrillation in Electrophysiological (EP) Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Heidelberg University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 235/04
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2006-10-12 (Estimated); Status verified 2004-11

CONDITIONS: Ventricular Fibrillation; Ventricular Tachycardia
Keywords: cerebral circulation
MeSH Terms: conditions — Ventricular Fibrillation; Tachycardia, Ventricular | interventions — Electroencephalography

INTERVENTIONS:
Device: EEG

SUMMARY:
In this study, changes in electroencephalogram (EEG) and the hemodynamic state during ventricular fibrillation or induced ventricular tachycardia are investigated.

DETAILED DESCRIPTION:
Patients with a high risk of malignant tachyarrhythmia are routinely investigated by programmed electrophysiological study (EPS). To investigate the hemodynamic effects of ventricular arrhythmia to cerebral circulation an EEG and transcranial ultrasound are conducted simultaneously during the EPS. Before and after the EPS a neuropsychological test and an investigation of a specific blood sample (Neuron Specific Enolase, NSE) is done.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Positive agreement
* EPS for primary and secondary prophylaxis of a malignant ventricular tachyarrhythmia:

  * primary prophylaxis: Brugada syndrome, long QT syndrome, cardiomyopathy, short QT syndrome
  * secondary prophylaxis: Multicenter Automatic Defibrillator Implantation Trial (MADIT) criteria, syncope, documented ventricular tachycardia

Exclusion Criteria:

* Severe neurological deficit
* Cardiopulmonary resuscitation

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 30

CONTACTS AND LOCATIONS:
Overall Officials: Martin Borggrefe, Prof., MD, Study Director — I.Medizinische Klinik, Universitätsklinikum Mannheim; M Hennerici, Prof., MD, Study Director — Neurologische Klinik Universitätsklinikum Mannheim
Locations (1):
- Fakultät für Klinische Medizin Mannheim Universitätsklinikum Mannheim der Ruprecht-Karls-Universität Heidelberg, Mannheim, Germany